CLINICAL TRIAL: NCT01800292
Title: Echo Study - Characterization of LV Strain Patterns in Patients With Mildly Elevated PCWP and Pulmonary Hypertension
Brief Title: Characterization of LV Strain Patterns in Mildly Elevated PCWP and PAH.
Acronym: LV strain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Aiden Abidov, Associate Professor, Medicine and Radiology, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-0006-01; 986-12 (Other: University Medical Center Site Review Authority)
Record Dates: First submitted 2013-02-22; First posted 2013-02-27 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension, Pulmonary Artery; Ventricular Dysfunction, Left
Keywords: Pulmonary Artery Hypertension; pulmonary capillary wedge pressure; sildenafil; echocardiography; left ventricular longitudinal wall strain; strain rate pre and post medical therapy; speckle tracking
MeSH Terms: conditions — Hypertension; Ventricular Dysfunction, Left; Familial Primary Pulmonary Hypertension | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sildenafil therapy (Experimental): Subjects will have 2D-Echocardiogram measuring left ventricular strain and strain rate using speckle tracking techniques, have 6 minute walk test, World Health Organization functional class (I-IV)assignment, and BNP lab result at baseline and at 3 months. Subjects will be started on sildenafil at 20 mg by mouth three times per day at the baseline visit. Each individual will serve as his/her own control.
  Interventions: Drug: sildenafil

INTERVENTIONS:
Drug: sildenafil — Subjects will be started on sildenafil at 20 mg PO TID at the baseline visit. Each individual will serve as his/her own control. Subjects will be evaluated at 3 months, with participation completed at that time.
  Other Names: Revatio; compound UK-92,480; Patent 5,250,534; sildenafil citrate; NDA 22-473; C22H30N6O4S.C6H8O7; C28H38N6O11S

SUMMARY:
The purpose of this study is to determine if patients with pulmonary hypertension and mildly elevated heart pressure known as PCWP will exhibit different patterns on echocardiography and that these patterns will predict treatment response to sildenafil, a drug given for this condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with New York Heart Association/World Health Organization(NYHA/WHO)functional class II-III
* Patients with mean pulmonary artery pressure >25 mmHg, pulmonary capillary wedge pressure >15 mmHg ≤18, and pulmonary vascular resistance >3 wood units
* Age >18 and <80
* Stable on antihypertensives and diuretics>3 months
* No evidence of active ischemic heart disease
* 6 minute walk distance >150 meters and <450 meters

Exclusion Criteria:

* - Left ventricular ejection fraction <50%
* Patients with significant restrictive lung disease (FVC<60% predicted) and/or significant obstructive lung disease (FEV1 <55% predicted) within 1 year of enrollment
* Poorly interpretable grey scale echocardiographic images
* Contraindications to right heart catheterization
* Nitroglycerin therapy
* Moderate-severe aortic and mitral valve abnormality
* Contraindications to submaximal exercise testing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
exercise capacity not on/on sildenafil therapy | 3 months
  Subjects will have 6 minute walk testing prior to sildenafil therapy and 3 months post-initiation of sildenafil therapy. Improvement in submaximal exercise capacity on sildenafil therapy is defined as ≥ 30 M increase in 6 minute walk testing.

SECONDARY OUTCOMES:
Echo parameters:left ventricular septal and lateral wall longitudinal strain and strain rate, RV strain and strain rate, and LV lateral wall/septal strain and strain rate | 3 months
  Echo parameters will be collected pre-therapy vs 3 months on sildenafil therapy. Changes in ventricular wall motion will be documented with left ventricular (LV) septal and lateral wall longitudinal strain and strain rate, right ventricular strain and strain rate, and LV lateral wall/septal strain and strain rate utilizing speckle tracking techniques values determined by 2D-Echo.

OTHER OUTCOMES:
World Health Organization functional class | 3 months
  World Health Organization functional class (I-IV) will be determined at baseline and at 3 months
BNP (brain natriuretic peptide) | 3 months
  Blood will be collected to get BNP (brain natriuretic peptide)lab result at baseline and at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Aiden Abidov, MD, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Medical Center, Tucson, Arizona, United States